CLINICAL TRIAL: NCT02228447
Title: Healthy Habits, Healthy Girls: a Intervention Program for Adolescent Girls From Disadvantaged Backgrounds
Brief Title: Healthy Habits, Healthy Girls Preventing Unhealthy Weight Gain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Sonia Tucunduva Philippi, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FSP_14
Record Dates: First submitted 2014-08-25; First posted 2014-08-29 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Overweight; Obesity
Keywords: Adolescent; Randomized controlled trial; Eating behavior; Physical Activity; Sedentary lifestyle
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention group (No Intervention): The control group will not receive any intervention during the one year of this study. Only the baseline, 6-12 months assessments (anthropometrics, PA, dietary intake, social cognitive mediators and sedentary behaviors). To prevent compensatory rivalry and resentful demoralization, the control school will be provided with a condensed version of the following 12-month assessments. The condensed version of the program will include the professional learning workshops for intervention schools and the intervention materials (i.e., nutrition and PA handbooks and PA leadership handbook).
- Healthy habits, healthy girls group (Experimental): The intervention group will receive a 6-month multicomponent intervention (i.e., enhanced physical education classes; interactive seminars; nutrition workshops; text messages; and parents newsletters) and materials (i.e., nutrition and PA handbooks; cooking books; Choreographies CDs and PA leadership handbook).
  Interventions: Behavioral: Healthy Habits, Healthy Girls Group

INTERVENTIONS:
Behavioral: Healthy Habits, Healthy Girls Group — The intervention group will receive a 6-month multicomponent intervention (i.e., enhanced physical education classes; interactive seminars; nutrition workshops; text messages; and parents newsletters) and materials (i.e., nutrition and PA handbooks; cooking books; Choreographies CDs and PA leadership handbook).
  Arms: Healthy habits, healthy girls group

SUMMARY:
The purpose of this study is to evaluate the impact of a multicomponent school-based intervention based on Bandura's Social Cognitive Theory targeting healthy eating and physical activity for high school adolescent girls from low-income communities in the city of São Paulo, Brazil.

DETAILED DESCRIPTION:
The "Healthy Habits, Healthy Girls" is a 6-month multi-component school-based intervention developed in reference to Social Cognitive Theory and includes: (1) enhanced physical education classes (2x/week and delivered by a Physical Education teacher), (2) break/lunch-time physical activity sessions (the participating girls will encourage younger girls to make Physical Activity during break and/or lunch-time. This session will only happen after 3 months of enhanced Physical Education classes, so the girls will be able to pass their knowledge for the others), (3) Nutrition and Physical Activity handbooks with 10 health messages (lessons to be done at home and their family); (4) 4 Parent newsletters; (5) Food and Physical Activity diaries for self-monitoring; (6) text-messages using a group application for more interaction and social support; and (7) 10 weekly Nutrition and Physical Activity key messages (delivered by a Nutrition and Dietetics Bachelor degree and/or Physical Education teacher during break). The intervention will be evaluated using a randomised controlled trial in 10 public schools in the city of São Paulo, Brazil (5 control and 5 intervention) and based on the 10 weekly key messages: (1) eat fruit and vegetables daily; (2) Do Physical Activity respecting your limits; (3) Eat a healthy breakfast every day; (4) Do Physical Activity with your family and friends; (5) Control the portion size you eat during meals - and sit while you are eating; (6) Reduce your sitting time during school break, after the school period and on the weekends; (7) Have less "junk food" for meals/snacks and munch less; (8) Identify the excuses for not practicing PA; (9) Drink water and substitute sodas and artificial juices for water, homemade natural fruit juices and coconut water, and; (10)Make family meals.

ELIGIBILITY:
Inclusion Criteria:

- Adolescent girls from low-income backgrounds enrolled in high schools of the city of São Paulo, Brazil.

Exclusion Criteria:

* Adolescent boys
* Adolescents from middle and high income backgrounds
* Pregnant

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 244 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 1 year
  Weight will be measured to the nearest 0.1kg without shoes, in light clothes using a portable digital scale and height was recorded to the nearest 0.1cm using a portable stadiometer. BMI was calculated using the standard equation (weight [kg]/height [m2]) and BMI z-score was calculated using the "LMS" method

SECONDARY OUTCOMES:
Dietary intake | 1 year
  Dietary intake was assessed a 49-item semi-quantitative food-frequency questionnaire (FFQ) Subjects were asked about their consumption over the previous 12-months. The frequency options ranged from "Never" to "at least twice a day" for all the items.
Physical activity level | 1 year
  PA was assessed using a brief PA questionnaire that aims to evaluate the PA frequency and intensity realized in one week. The subjects should inform the number of times of light-to-vigorous intensity PA practiced for at least 30 minutes during a period of seven days (i.e., week and weekends).
Sedentary behaviors | 1 year
  The subjects reported the time spent during the weekdays (Monday through Friday) and weekends (Saturday and Sunday) in the following activities: watching television/videos/DVDs, using the computer for leisure activities (games and social networks), using telephone and studying, reading or doing homework.
Physical activity social-cognitive mediators | 1 year
  Social cognitive scales for dietary and PA behaviors based on constructs from Social Cognitive Theory were adapted and designed for the study. Participants will complete PA scales for the following constructs: self-efficacy, intentions, family and friends support, environment perceptions (situation), behavioral strategies (self-control), outcome expectations (perceived benefits) and outcome expectancies (valued placed on benefits).
Dietary social cognitive mediators | 1 year
  Social cognitive scales for dietary behaviors based on constructs from Social Cognitive Theory were adapted and designed for the study. Participants will complete dietary scales for the following constructs: self-efficacy, intentions, family and friends support, environment perceptions (situation), behavioral strategies (self-control), outcome expectations (perceived benefits) and outcome expectancies (valued placed on benefits)
Waist circunference | 1 year
  waist circumference will be measured to the nearest 0.1cm against the skin using a non-extensible steel tape in line with the umbilicus.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Tucunduva Philippi, PhD, Study Chair — School of Public Health University of São Paulo; Ana Carolina Barco Leme, Master, Principal Investigator — School of Public Health, University of São Paulo
Locations (1):
- School of Public Health, University of São Paulo, São Paulo, São Paulo, Brazil